CLINICAL TRIAL: NCT01656226
Title: A Randomised Double-blind Parallel-group Study to Evaluate the Long-term Effects of Eryfotona AK-NMSC® Cream in the Treatment of Cancerization Field in Patients With Actinic Keratosis.
Brief Title: Long Term Efficacy and Safety of Eryfotona AK-NMSC® in Patients With Actinic Keratosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ISDIN (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISD-FPT-01-2012
Record Dates: First submitted 2012-07-24; First posted 2012-08-02 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2012-08

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratosis; AK
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eryfotona AK-NMSC® cream (Experimental)
  Interventions: Device: Eryfotona AK-NMSC® cream
- Sunscreen SPF 50+ (Other)
  Interventions: Other: Sunscreen SPF 50+

INTERVENTIONS:
Device: Eryfotona AK-NMSC® cream — Cream, to be applied according to COLIPA standard at 2 mg/cm² in head and neck, twice a day before exposing to sun light morning and around lunchtime (about 4-6 hours later), for up to 6 months.
  Arms: Eryfotona AK-NMSC® cream
Other: Sunscreen SPF 50+ — Cream, to be applied according to COLIPA standard at 2 mg/cm² in head and neck, twice a day before exposing to sun light morning and around lunchtime (about 4-6 hours later), for up to 6 months.
  Arms: Sunscreen SPF 50+

SUMMARY:
The purpose of this study is to assess the efficacy, safety and tolerability of Eryfotona AK-NMSC® topical application vs Sunscreen on cancerization field of actinic keratosis patients after 6 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Current diagnosis of AK, with ≥4 lesions located in the same anatomical district (within a contiguous 50 cm2 area on the face, bold scalp or forehead);
2. Female or male >18 years of age;
3. Skin type I or II according to Fitzpatrick;
4. Patient has confirmed his/her willingness to participate in this study;.

Exclusion Criteria:

1. Topical drug therapy for AK within the past 3 months or for photoaging in the last 6 months, or had lesion-directed therapy within 2 cm2 of the selected AK area during the previous month;
2. Suitable for surgical, photodynamic or any other topical treatment in the next 6 months;
3. Subjects who suffer/ had suffered from skin cancer or show an early stage of skin cancer or have a genetic predisposition for skin cancer;
4. Other skin disease that requires treatment with other medications in the treatment area or in the distance of 3 cm;
5. Immunosuppression or current treatment for cancer;
6. Clinically unstable medical condition;
7. High risk group for HIV infection or presentation of other infectious diseases
8. Presentation of contact allergies or allergies to compounds of the test substances;
9. Smoker (more than forty cigarettes per day) or heavy drinker (more than three standard drinks per day);
10. Psychiatric disease that may interfere with follow up of study procedures;
11. Participation in other clinical trials up to 30 days prior to day 1 of the study
12. Prior treatment with study medication in the area to be treated;
13. Considered by the investigator, for any other reason, to be an unsuitable candidate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with partial clearance of AK lesions | 6 months
  Comparison between treatment groups at the end of the treatment period

SECONDARY OUTCOMES:
Percentage of patients with clearance and improvement of AK lesions | 6 months
  Comparison between treatment groups at the end of the treatment period
Total number of AK lesions in the treated area (including all lesions present at baseline as well as subclinical lesions which appeared during therapy) | 6 months
  Comparison between treatment groups at the end of the treatment period
Percentage of patients with improvement (clinical and dermoscopic assessment) of the target area as for the erythema, scaling, pigmentation and follicular plugs | 6 months
  Comparison between treatment groups at the end of the treatment period
Percentage of patients with changes in the Investigator Global Improvement Index | 6 months
  Comparison between treatment groups at the end of the treatment period
Percentage of patients with changes in Baseline Severity Index (BSI) | 6 months
  Comparison between treatment groups at the end of the treatment period
Percentage of patients with improvement in the target AK lesion by using RCM score. | 6 months
  Comparison between treatment groups at the end of the treatment period
Percentage of patients with improvement in the "cancerization filed" by RCM score | 6 months
  Comparison between treatment groups at the end of the treatment period Validation of a new RCM score
Percentage of patients compliant to treatment | 6 months
  Comparison between treatment groups at the end of the treatment period
Percentage of patients which report satisfaction to local tolerability | 6 months
  Comparison between treatment groups over time and at the end of the treatment period
Number of patients with AEs and local AEs (skin reactions) | 6 months
  Comparison between treatment groups over time and at the end of the treatment period
Percentage of patients which report satisfaction to treatment | 6 months
  Comparison between treatment groups at the end of the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Giuseppe Argenziano,, MD, PhD, Principal Investigator — Dermatology Unit, Medical Department /Arcispedale Santa Maria Nuova /Reggio Emilia, Italy
Locations (1):
- Dermatology Unit, Medical Department Arcispedale Santa Maria Nuova, Reggio Emilia, Italy